CLINICAL TRIAL: NCT04737005
Title: Evaluation of Marginal and Internal Adaptation and Clinical Performance of Endo-crowns Fabricated From Nano-ceramic Hybrid and Lithium Di-silicate Ceramic Materials (A Randomized Controlled Clinical Trial)
Brief Title: Evaluation of Marginal, Internal Adaptation and Clinical Performance of Endo-crowns Fabricated From Nano Hybrid and Lithium Di-silicate Ceramic Materials.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Salahel-din Abdel-azim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191020
Record Dates: First submitted 2021-01-26; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Clinical Fit and Clinical Performance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano-ceramic hybrid (Grandio Blocs) Endo-crown. (Other): Nano-ceramic hybrid ( intervention)
  Interventions: Procedure: Nano-ceramic hybrid (Grandio Blocs) Endo-crown
- Lithium di-silicate Ceramic (E.max CAD blocks) Endo-crown (Active Comparator): Lithium di-silicate Ceramic ( Control)
  Interventions: Procedure: Nano-ceramic hybrid (Grandio Blocs) Endo-crown

INTERVENTIONS:
Procedure: Nano-ceramic hybrid (Grandio Blocs) Endo-crown — Nano-ceramic hybrid

SUMMARY:
Evaluation of the marginal and internal adaptation using silicon replica technique, which will be measured by digital microscope and clinical Performance using modified USPHS scoring system of Endo-crowns fabricated from Nano-ceramic Hybrid and Lithium di-silicate ceramic materials.

DETAILED DESCRIPTION:
Evaluation of the marginal and internal adaptation using silicon replica technique, which will be measured by digital microscope and clinical Performance using modified USPHS scoring system of Endo-crowns fabricated from Nano-ceramic Hybrid and Lithium di-silicate ceramic materials.

Primary outcome: Marginal gap of the two groups will be measured using Silicon replica technique, Each replica will be sectioned bucco-lingually and mesio-distally into four segments named (MB, DB, ML, DL) and each segment has five reference points assigned at different positions, An overall of twenty reference points will be measured in each replica sample using a digital microscope.

Secondary outcome:

* Internal gap of the two groups will be measured using Silicon replica technique, which will be measured by digital microscope.
* Clinical Performance of the two groups will be evaluated using modified USPHS scoring system. (Color match, Marginal discoloration, Surface texture and Gross fracture)

ELIGIBILITY:
Inclusion Criteria:

* From 18-50 years old, be able to read and sign the informed consent document.
* Have no active periodontal or pulpal diseases, have teeth with good restorations.
* Psychologically and physically able to withstand conventional dental procedures.
* Patients planned for a single coverage restoration in the posterior area.
* Able to return for follow-up examinations and evaluation.
* Patients have root apex of molar without evident damage and no root fracture.
* Good oral hygiene habits.
* Have a complete root canal therapy molar necessitating an Endo-crown restoration.

Exclusion Criteria:

* Patient less than 18 or more than 50 years
* Patients with severe clenching or bruxism.
* Patient with active resistant periodontal diseases
* Patients with poor oral hygiene and uncooperative patients
* Pregnant women
* Patients in the growth stage with partially erupted teeth
* Psychiatric problems or unrealistic expectations
* Patients with inadequate or low quality endodontic treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Marginal and internal gap evaluation | 1 year
  marginal and internal gap will be evaluated by silicon replica technique, each replica will be sectioned into four segments named (MB, DB, ML, DL) and each segment had five reference points assigned at different positions, an overall of twenty reference points will be measured in each replica sample using a digital microscope. The measuring unit by microns

SECONDARY OUTCOMES:
clinical performance(Color match, Marginal discoloration, Surface texture and Gross fracture) | 1 year
  Clinical performance will be measured by modified USPHS criteria and the measuring unit by Alpha (A), Bravo (B) and Charlie (C)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR